CLINICAL TRIAL: NCT02490735
Title: A Randomized Controlled Study of Cytokine-induced Killer Cells (CIK) Treatment in Patients With Staging Ⅰ-Ⅲ of Esophageal Carcinoma
Brief Title: CIK in Treating Patients With Esophageal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESCC-CZYY-01
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No-CIK (No Intervention): After accepting chemotherapy, patients will regularly follow up.
- CIK (Experimental): After accepting chemotherapy, patients will receive at least 3 cycles of Cytokine-induced Killer Cells treatment per year
  Interventions: Biological: Cytokine-induced Killer Cells

INTERVENTIONS:
Biological: Cytokine-induced Killer Cells — chemotherapy plus 3 cycles of Cytokine-induced Killer Cells(CIK) treatment
  Other Names: CIK
  Arms: CIK

SUMMARY:
Chemotherapy is the main treatment method for patients with Esophageal Cancer. However, Relapse remains the major cause of treatment failure.Biological therapies such as CIK stimulate the immune system and stop tumor cells from growing. A series of studies reported that cytokine-induced killer cells (CIK) have a broad anti-tumor spectrum. The investigators suppose that CIK will improve the prognosis. Combining chemotherapy with biological therapy may kill more tumor cells. In this study, the patients will be treated with CIK cells after chemotherapy. The purpose of this study is to evaluate the efficacy of CIK for Esophageal Cancer.

DETAILED DESCRIPTION:
About 2000 patients with staging I-III of Esophageal Cancer, after accepting chemotherapy, will be randomly divided into group A (receive CIK treatment) or group B (just regularly follow up), and the randomize ratio will be 1:1. Patients in group A will receive 3 cycles of CIK cells treatment (every 12 weeks). Patients in group B will have no anti-tumor therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients histologically confirmed esophageal carcinoma;
* Patients with staging I-III of esophageal carcinoma;
* Patients who had completed chemotherapy;
* Patients who have a life expectancy of at least 12 weeks;
* Eastern Cooperative Oncology Group (ECOG) performance status was 0-1;
* The bone marrow functioned normally (WBC>4.0×10^9/L, Hb>120 g/L, Platelet(PLT)>100×10^9/L);
* The ECG results were normal, and the liver and kidney were functional.

Exclusion Criteria:

* Patients who had distant metastases by imaging studies;
* Patients with uncontrolled infection; underlying disease that was severe or life-threatening;
* Patients who were lactating;
* ECOG perform status ≥ 2;
* Patients who are suffering from auto immune diseases or patients who need to accept glucocorticoid treatment;
* Patients who are pregnant or nursing;
* Patients with active tuberculosis (highly positive skin tests allowed if no active disease);
* Patients with disease that would preclude general anesthesia;
* Patients with active intractable or uncontrollable infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2015-08; Primary Completion 2040-08 (Estimated); Study Completion 2042-08 (Estimated)

PRIMARY OUTCOMES:
progression-free survival(PFS) | 1 month

SECONDARY OUTCOMES:
overall survival(OS) | 1 month

OTHER OUTCOMES:
Stage at diagnosis | 1 month
  Tumor Node Metastasis (TNM) stage, Tumor:CIS,T1,T2,T3,T4 according to the depth of tumor invasion. Lymph node involvement: N0,N1,N2. Metastasis: M0,M1